CLINICAL TRIAL: NCT05819996
Title: Addressing Tetrachloroethylene Exposure in an Impacted Community: Residents' Concerns, Neurotoxic Effects, and Exposure Reduction
Brief Title: Addressing Tetrachloroethylene Exposure in an Impacted Community
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: University of Illinois at Chicago (Other); Indiana University School of Medicine (Other); Mackey Children's Cancer Foundation (Unknown)
Responsible Party: Principal Investigator, Sa Liu, Assistant Prof., Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20211507
Record Dates: First submitted 2022-12-05; First posted 2023-04-19 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-05

CONDITIONS: Vapors; Inhalation; Cancer; Volatile Organic Compounds
Keywords: Tetrachloroethylene; Trichloroethylene; PCE; TCE; Community environmental contamination; Chlorinated volatile organic compounds
MeSH Terms: conditions — Respiratory Aspiration; Neoplasms

STUDY DESIGN:
Intervention Model Description: An educational campaign targeting the community
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Martinsville Residents (Other): Residents of Martinsville, Indiana, will receive educational campaign promoting participation in environmental testing
  Interventions: Behavioral: Environmental educational campaign

INTERVENTIONS:
Behavioral: Environmental educational campaign — Educational campaign will be conducted to promote participation in indoor air testing.

SUMMARY:
Groundwater in Martinsville, IN, is contaminated by volatile organic compounds (VOCs), tetrachloroethylene (PCE) and trichloroethylene (TCE). Indoor air in some residential and commercial buildings is also contaminated with PCE and TCE. This study is being conducted to better understand the impact of low-level exposures to these compounds on community members' health. Data collected in this study will be used to help the community identify a course of action.

DETAILED DESCRIPTION:
Martinsville, IN, is a community of 11,000 people that overlays four groundwater contamination sites, including a U.S. Environmental Protection Agency (EPA)-designated Superfund site. The total area of groundwater contamination is over 60 acres and lies within a single aquifer. The contaminates are chlorinated volatile organic compounds (VOCs), primarily tetrachloroethylene (PCE) and trichloroethylene (TCE). These contaminants are thought to originate from several dry cleaning and metal degreasing operations. An activated carbon filtration system has been in operation since 2005 to remove PCE and chlorinated VOCs from the municipal water, which now meets EPA drinking water standards. However, a recent report from the Agency for Toxic Substances and Disease Registry concludes that people's health may be harmed by breathing indoor air contaminated via vapor intrusion, the migration of volatile compounds from contaminated groundwater and soil into buildings above. The long-term goal of this research is to understand how PCE exposure in communities affects health and to empower community members' participation in environmental health decision-making. In this project researchers will work with the community of Martinsville, IN to:

1. Determine the extent and exposure levels to the contaminants by measuring the contamination in residents and at their homes.
2. Assess the community's concern and perceptions about the contamination and associated health risks.
3. Study the impact of the contaminants on visual and neurocognitive functions.
4. Compare cancer rates in Martinsville to county and state rates.

The above information will help researchers and community partners co-design a targeted educational campaign to reduce community members' exposure to the contaminants.

ELIGIBILITY:
Inclusion Criteria:

* Residents of Martinsville, Indiana
* 18 years or older

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in concerns about environmental chemical contamination in Martinsville. | For Measure 1a, Time frame is from year 1 to year 3; for Measure 1b, Time frame is from year 1 to year 5.
  This measure is based on the differences between the percentage of "Yes" responses to a close-ended, not scaled question at 3 different time points, administered via repeated surveys to the same sample of respondents.
  Are participants concerned about environmental chemical contamination in Martinsville? Yes / Somewhat / No / Refuse
  1a. Changes in concerns about environmental chemical contamination in Martinsville from Year 1 to Year 3. This is based on the differences in percentage of yes responses to this question in surveys administered in Year 1 (Main survey, baseline) and Year 3 (online survey administered at the beginning of Year 3).
  1b. Changes in concerns about environmental chemical contamination in Martinsville from Year 1 to Year 5. This is based on the differences in percentage of yes responses to this question in surveys administered in Year 1 (Main survey, baseline) and Year 5 (Online survey, post intervention).
Changes in awareness of possible exposure to chemicals from soil or groundwater in Martinsville. | For Measure 2a, Time frame is from year 1 to year 3; for Measure 2b, Time frame is from year 1 to year 5.
  This measure is based on the differences between the percentage of "Yes" responses to a close-ended, not scaled question at 3 different time points, administered via repeated surveys to the same sample of respondents.
  Are participants aware of possible exposure to chemicals from soil or groundwater in Martinsville? Yes / No / Refuse
  2a. Changes in awareness of possible exposure to chemicals from soil or groundwater in Martinsville from Year 1 to Year 3. This is based on the differences in percentage of yes responses to this question in surveys administered in Year 1 (Main survey, baseline) and Year 3 (Online survey administered at the beginning of Year 3).
  2b. Changes in awareness of available resources for exposure reduction from Year 1 to Year 5. This is based on the differences in surveys administered in Year 1 (Main survey, baseline) and Year 5 (Online survey, post intervention)
Change in willingness to have respondent's homes tested for chemical contamination from contaminated soil or groundwater. | For Measure 3a, Time frame is from year 1 to year 3; for Measure 3b, Time frame is from year 1 to year 5.
  This measure is based on the difference between the percentage of "Yes" responses to a close-ended, not scaled question at 3 different time points, administered via repeated surveys to the same sample of respondents.
  Are participants willing to have their home tested for chemical contamination from contaminated soil or groundwater? Yes / No / Refuse / Don't know
  3a. Changes in willingness to have respondents' homes tested for the chemical contamination from Year 1 to Year 3. This is based on the differences in percentage of yes responses to this question in surveys administered in Year 1 (Main survey, baseline) and Year 3 (Online survey at the beginning of Year 3)
  3b. Changes in willingness to have respondents' homes tested for the chemical contamination from Year 1 to Year 5. This is based on the differences in differences in percentage of yes responses to this question in surveys administered in Year 1 (Main survey, baseline) and Year 5 (Online survey, post intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Sa Liu, MPH, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No